CLINICAL TRIAL: NCT01949883
Title: A Phase 1 Study of CPI-0610, a Small Molecule Inhibitor of BET (Bromodomain and Extra-terminal) Proteins, in Patients With Progressive Lymphoma
Brief Title: A Phase 1 Study Evaluating CPI-0610 in Patients With Progressive Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Constellation Pharmaceuticals (Industry)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0610-01
Record Dates: First submitted 2013-09-10; First posted 2013-09-25 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Lymphoma
Keywords: Phase 1; Oncology; BET Inhibitor
MeSH Terms: conditions — Lymphoma; Neoplasms | interventions — CPI-0610

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CPI-0610 (Experimental)
  Interventions: Drug: CPI-0610

INTERVENTIONS:
Drug: CPI-0610

SUMMARY:
First in human, open-label, sequential dose escalation and expansion study of CPI-0610 in patients with progressive lymphoma. CPI-0610 is a small molecule inhibitor of bromodomain and extra-terminal (BET) proteins.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged ≥ 18 years)
* Histologically confirmed diagnosis of a non-Hodgkin or Hodgkin lymphoma that has progressed in spite of prior treatment, and for which additional effective standard therapy is not available
* Patients may have either measurable or non-measurable disease, but in all cases eligible patients must have disease that can be clinically evaluated for improvement or progression
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Adequate hematological, renal, hepatic, and coagulation laboratory assessments
* Written informed consent to participate in this study before the performance of any study-related procedure

Exclusion Criteria:

* A primary lymphoma of the central nervous system (CNS) or known lymphomatous involvement of the CNS. CNS imaging and cerebrospinal fluid sampling are not mandatory in the absence of a clinical suspicion of lymphomatous involvement of the CNS.
* Current infection with HIV, Hepatitis B or Hepatitis C. Patients will have serologic testing performed during screening for HIV and Hepatitis B and C. Any serologic results suggestive of an ongoing viral infection will be further investigated as necessary to clarify the patient's status.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of CPI-0610, including any unresolved nausea, vomiting, or diarrhea that is CTCAE grade >1.
* Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

  * Acute myocardial infarction or angina pectoris ≤ 6 months prior to starting study drug
  * Serum cardiac troponin (cTn) level ≥ 99% percentile of the upper reference limit
  * QTcF > 470 msec on the screening ECG
  * Left ventricular ejection fraction (LVEF) < 40%
* Uncontrolled cardiac arrhythmia (patients with rate-controlled atrial fibrillation are not excluded.)
* Any other concurrent severe and/or uncontrolled concomitant medical condition that could compromise participation in the study (e.g., clinically significant pulmonary disease, clinically significant neurological disorder, active or uncontrolled infection)
* Systemic anti-cancer treatment or radiotherapy less than 2 weeks before the first dose of CPI-0610
* Radioimmunotherapy (e.g., 131I-tositumomab, 90Y-ibritumomab tiuxetan) less than 6 weeks before the first dose of CPI-0610
* Treatment with an investigational small molecule less than 2 weeks before the first dose of CPI-0610. In addition, the first dose of CPI-0610 should not occur before a period equal to or greater than 5 half-lives of the small molecule investigational agent has elapsed.
* Treatment with a therapeutic antibody less than 4 weeks before the first dose of CPI-0610. A minimum 2-week period between the last treatment with a therapeutic antibody and the first dose of CPI-0610 may be permitted in patients with rapidly progressive or aggressive subtypes of lymphoma following discussion with the medical monitor.
* Treatment with medications that are known to be strong inhibitors or inducers of CYP450 enzymes.
* Treatment with medications that are known to carry a risk of Torsades de Pointes.
* Immunosuppressive treatment that cannot be discontinued both prior to study entry and for the duration of the study. Oral prednisone at a dose of 10 mg or less per day is allowed, as are other oral corticosteroids given at glucocorticoid-equivalent doses. Topical, nasal and inhaled corticosteroids are also allowed.
* Pregnant or lactating women
* Women of child-bearing potential and men with reproductive potential, if they are unwilling to use adequate contraception while on study therapy and for 3 months thereafter
* Patients unwilling or unable to comply with this study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-09-05 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Frequency of dose-limiting toxicities (DLTs) associated with CPI-0610 administration during the first cycle (first 21 days) of treatment | DLTs asessed during Cycle 1 (first 21 days on study)

SECONDARY OUTCOMES:
Safety and tolerability of CPI-0610 as assessed by: frequency of adverse events and serious adverse events; changes in hematology and clinical chemistry values; changes in physical examination, vital signs, electrocardiogram, ECHO and ECOG score | Assessed from Day 1 of Cycle 1 through 30 days after patient's last dose of study drug
Pharmacokinetic parameters of CPI-0610: AUC(0-t), AUC(0-inf), AUCtau,ss, Tmax, Cmax, Ctrough, T1/2, Vd/F, CL/F | Assessed during cycle 1 (first 21 days on study); and on cycle 2, day 1
Pharmacodynamic effects of CPI-0610: Changes in the expression of MYC and other genes in tumor tissue; changes in cellular proliferation and in the extent of apoptosis; changes in tumor metabolism | Assessed during cycle 1 (first 21 days on study); and on cycle 2, day 1
Changes in the expression of a set of genes in peripheral blood mononuclear cells (PBMCs) that are sensitive to BET inhibition | Assessed during cycle 1 (first 21 days on study)
Anti-lymphoma activity associated with CPI-0610 treatment | After every 2 cycles of treatment for the first 6 cycles, and after every 4 cycles thereafter; assessed up to approximately 12 months

REFERENCES:
- [Derived] Blum KA, Supko JG, Maris MB, Flinn IW, Goy A, Younes A, Bobba S, Senderowicz AM, Efuni S, Rippley R, Colak G, Trojer P, Abramson JS. A Phase I Study of Pelabresib (CPI-0610), a Small-Molecule Inhibitor of BET Proteins, in Patients with Relapsed or Refractory Lymphoma. Cancer Res Commun. 2022 Aug 11;2(8):795-805. doi: 10.1158/2767-9764.CRC-22-0060. eCollection 2022 Aug. PMID 36923307